CLINICAL TRIAL: NCT02600364
Title: Prospective, Multicenter, Single Arm Post Market Clinical Follow-Up Study to Assess Safety and Effectiveness of the p64 Flow Modulation Device
Brief Title: Diversion-p64 Post Market Clinical Follow-Up Study to Assess Safety and Effectiveness of the p64 Flow Modulation Device
Status: Completed | Type: Observational
Sponsor: Phenox GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: DP64/BO1507
Record Dates: First submitted 2015-11-04; First posted 2015-11-09 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Intracranial Aneurysm
Keywords: Aneurysm; intracerebral; stroke; p64
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm; Stroke; X-Linked Combined Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess safety and effectiveness of the p64 Flow Modulation Device.

DETAILED DESCRIPTION:
Title: Diversion-p64. Device: p64 Flow Modulation Device. Study design: Prospective, multicenter, single arm Post Market Clinical Follow-Up Study.

Purpose: To assess safety and effectiveness of p64. Study duration: 48 months. Sample Size: 400 patients. Number of sites: > 20. Follow-up intervals: Two independent follow-ups (after 3-6 and 7-12 months) according to site specific standard.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18
2. Patient harbours either one saccular or one dissecting or one blisterlike or one fusiform intracerebral aneurysm or one intracerebral segmental disease, in the anterior circulation for which the indication for p64 treatment is given
3. Patient or legal representative provides written informed consent verifying that he/she consents to the use of his/her data (according to the data protection laws)

Exclusion Criteria

1. Aneurysms of the posterior circulation
2. Imaging evidence of bifurcation aneurysms
3. Imaging evidence of dissections
4. Imaging evidence of fistulae
5. Imaging evidence of arteriovenous malformations
6. Patient is harbouring another aneurysm that has to be treated within six months after first procedure
7. Known allergy to study medication, e.g. ASA, Clopidogrel, Heparin or contrast media
8. Confirmation of positive pregnancy test according to site specific standard of care (e.g. test, verbal communication)
9. Current involvement in another study or trial
10. Parent vessel treated with other Flow Diverters than p64 during intervention and re-treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this non-interventional study are patients with ruptured or unruptured aneurysms and segmental diseases in the anterior circulation. Patients can be included in the study if they meet all of the inclusion and none of the exclusion criteria and have provided written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change in the rate of complete occlusion | immediately after treatment, an expected average of 1 hour; to 12 months
  Rate of complete aneurysm occlusion is assessed immediately after treatment (an expected average of 1 hour) and at both follow-up visits (3-6 months and 7-12 months). The change is assesed.
Change of frequency of major stroke (ischemic or hemorrhagic) or neurological death related to the treatment of the target aneurysm | immediately after treatment, an expected average of 1 hour; to 12 months
  Frequency of major stroke (ischemic or hemorrhagic) or neurological death is assessed immediately after treatment (an expected average of 1 hour) and at both follow-up visits (3-6 months and 7-12 months). The change is assesed.

SECONDARY OUTCOMES:
Intra-procedural technical complications | during treatment, an expected average of 1 hour
  p64 placed in the desired location Correct opening of p64 (markers fully deployed) at the end of the procedure Ability to detach p64 at the end of the procedure
Change of Angiographic results | immediately after treatment, an expected average of 1 hour; to 12 months
  Change in both Rate of re-growth (related rate of re-treatment) and Rate of recanalization (related rate of re-treatment) are assessed immediately after treatment (an expected average of 1 hour) and at both follow-up visits (3-6 months and 7-12 months).
Intra-procedural vascular complications | during treatment, an expected average of 1 hour
  Vessel perforation (e.g. with distal wire tip of p64, microcatheter) Target aneurysm perforation (e.g. with distal wire tip of p64, microcatheter) Thromboembolism Dissection of any access vessel Side branch occlusion
Post-procedural Complications | 3-6 and 7-12 months
  Parenchymal hemorrhage detected during the follow-up period Subarachnoid hemorrhage detected during the follow-up period Ischemic stroke detected on follow-up imaging Rupture of the target aneurysm detected during the follow-up period Rate of in-stent-stenosis detected during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Alain Bonafé, Prof. Dr., Principal Investigator — Hôpital Gui de Chauliac (CHU de Montpellier), Montpellier, France
Locations (26):
- Clínica La Sagrada Familia, Buenos Aires, Argentina
- Ziekenhuis Oost-Limburg, Genk, Belgium
- St. Ivan Rilski Hospital, Sofia, Bulgaria
- France (7):
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Hôpital Pierre Wertheimer, Bron
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Gui de Chauliac (CHU Montpellier), Montpellier
  - Hôpital Pitié Salpétrière, Paris
  - CHRU Hôpital Maison-Blanche, Reims
  - Hôpital Bretonneau (CHRU de Tours), Tours
- Germany (6):
  - Klinikum Augsburg, Augsburg
  - Klinikum Bremen-Mitte, Bremen
  - HELIOS Klinikum Erfurt, Erfurt
  - Knappschaftskrankenhaus Recklinghausen, Recklinghausen
  - Universitätsklinikum Regensburg, Regensburg
  - Klinikum Stuttgart Katharinenhospital, Stuttgart
- Italy (2):
  - Ospedale Bellaria Carlo Alberto Pizzardi, Bologna
  - IRCCS Istituto Clinico Humanitas, Rozzano
- Poland (2):
  - Regionalny Szpital Specjalistyczny, Grudziądz
  - Uniwersytecki Szpital Kliniczny we Wroclawiu, Wroclaw
- Life Memorial Hospital, Bucharest, Romania
- Russia (2):
  - NSI Burdenko, Moscow, Moscow
  - Federal Almazov North-West Medical Research Centre, Saint Petersburg
- United Kingdom (3):
  - Western General Hospital, Edinburgh
  - Leeds Teaching Hospitals NHS TRUST, Leeds
  - St George's Hospital, London

REFERENCES:
- See also: www.phenox.net — http://phenox.net/